CLINICAL TRIAL: NCT05338112
Title: Evaluation of the Relationship of Tzanck Smear Findings And Disease Activity In Patients With Pemphigus Vulgaris
Brief Title: Role of Tzanck Smear in Determining Pemphigus Vulgaris Disease Activity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Zeynep Arslan, Doctor of Medicine, Istanbul Medeniyet University
Other Study IDs: 10457119
Record Dates: First submitted 2022-04-07; First posted 2022-04-20 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-04

CONDITIONS: Pemphigus Vulgaris
Keywords: pemphigus vulgaris, Tzanck smear, disease activity, prognostic factor
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with active pemphigus lesions
  Interventions: Diagnostic Test: Tzanck smear

INTERVENTIONS:
Diagnostic Test: Tzanck smear — The Tzanck smear is gently taken with a sterile scalpel from the ground of erosion or bullous lesions of pemphigus vulgaris. The sample taken is examined by staining the slide.

SUMMARY:
Aim: Pemphigus vulgaris (PV) is a rare, life-threatening autoimmune bullous disease that can involve the skin and mucous membranes, characterized by intraepidermal bullae and eroded lesions caused by rupture of the bullae. The aim of this study is to research the relationship of the findings obtained with Tzanck smear, which is an inexpensive and easy method, with disease activity and its prognostic importance in the clinical course in PV patients.

Material and Methods: Pemphigus patients who visited to Goztepe Prof. Dr. Suleyman Yalcın City Hospital, Dermatology Clinic will be included in our study. Pemphigus disease area index (PDAI), Tzanck smear findings from the lesions and desmoglein levels during routine follow-up of patients with pemphigus vesicle/bulla/erosion will be evaluated. In the evaluation of Tzanck smear preparations, the entire slide will be scanned, acantholytic cell count performed and scored 1 to 4 accordingly (1 point: 1-3 cells, 2 points: 4-10 cells, 3 points:11-20, 4 points: >21 cells or cell clusters). Anti-desmoglein antibody levels will be analyzed by using enzyme-linked immunosorbent assay (ELISA) method.

ELIGIBILITY:
Inclusion Criteria:

* Clinical, histopathological and immunological diagnosis of pemphigus vulgaris
* Must be active bullae or erosion at any stage of the disease

Exclusion Criteria:

* Patients with uncertain diagnosis of pemphigus vulgaris
* Eroded lesions due to causes other than pemphigus vulgaris (such as herpes in the oral mucosa, candida infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with pemphigus vulgaris by clinical, histopathological and immunological methods.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
The number of acantholytic cells | 1or 2 months
  Tzanck smear slides will be entirely scanned, acantholytic cell count will be performed and scored 1 to 4 accordingly (1 point: 1-3 cells, 2 points: 4-10 cells, 3 points:11-20, 4 points: >21 cells or cell clusters).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes